CLINICAL TRIAL: NCT02431026
Title: Temperature Evaluation by MRI Thermometry During Cervical Cooling
Acronym: TEM-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Cryothermic Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Wolfson, MD, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TEM-C
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: induced mild hypothermia; cervical cooling collar; mri brain thermometry; MRI thermometry; rate-of-cooling; Excel Cryo Cooling Collar

ARMS (2):
- Cooling present (Experimental): Cooling pack activated before start of MRI scan for the condition "cooling present".
  Interventions: Device: Cooling pack activated Excel Cryo Cooling Collar
- No cooling present (No Intervention): Cooling pack will not be activated in the condition "no cooling present".

INTERVENTIONS:
Device: Cooling pack activated Excel Cryo Cooling Collar — Cooling pack will be activated before insertion into collar. The first cooling pack will be replaced 20 minutes later with a new, activated cooling pack.
  Arms: Cooling present

SUMMARY:
The American Heart Association (AHA) recommends cooling (inducing mild hypothermia) patients who were resuscitated following cardiac arrest but who remained comatose. Induced mild hypothermia is now the standard of care for post-resuscitation patients in the intensive care unit (ICU) setting. The use of cooling has recently moved to pre-hospital and emergency department (ED) application as more current studies show that early initiation of cooling significantly improves neurologic outcomes and survival rates instead of waiting until the patient arrives in the ICU to initiate cooling. In the pre-hospital setting chilled saline (4°C) and packing the body in ice have been the primary methods to initiate induced mild hypothermia The Excel Cryo Cooling System is a non-invasive cervical collar (C-collar) that provides cooling to the carotid arteries, the main blood supply to the brain, and allows for the rapid initiation of selective cerebral cooling. The investigators are planning to use MRI-thermometry to see how quickly the Excel Cryo Cooling Collar can drop brain temperature when applied by itself.

Healthy volunteers will be used for this study to provide important temperature data on the effectiveness of the Excel Cryo Cooling System. The investigators will be able to use the data from this project to further the current clinical research in induced mild hypothermia after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Understands the risks involved, as detailed in the informed consent
* No MRI risk factors

Exclusion Criteria:

* < 18 years of age & > 60 years of age
* Pregnant
* Any known medical problems that limit activity or decrease blood flow: underactive thyroid (hypothyroidism),poor nutrition, stroke, severe arthritis, Parkinson's disease, dementia, significant mental illness besides clinical depression, spinal cord injuries, recent serious burn, disorders that affect sensation in the extremities (e.g., diabetic neuropathy)dehydration, and any condition that limits activity or restrains the normal flow of blood.
* Taking any medications (except seasonal allergy medication, over-the-counter NSAIDs, acetaminophen, or contraceptives)
* Oral medications that inhibit the body's ability to respond to cold: Antidepressants, antipsychotics/neuroleptics, including phenothiazines, beta blockers, clonidine, meperidine, sedative-hypnotics.
* History of cardiac condition in a family member younger than 40 years
* Inability to fit in the MRI scanner (BMI > 30 kg/m2)
* MRI risk factors (e.g., claustrophobia, heart condition, metal implants, etc), as detailed in the MRI safety questionnaire Heart rate, blood pressure, respiratory rate, or temperature outside of acceptable ranges.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rate of cooling | 45 minutes
  MRI thermometry will be used to evaluate the rate of cooling
Time to drop subject temperature 0.8-3.0°C | 45 minutes
  Temperatures changes will be evaluated using MRI thermometry
Time to induced mild hypothermia threshold (34ºC) | 45 minutes
  Temperatures changes will be evaluated using MRI thermometry
Differences and similarities of inducing mild hypothermia with the Excel Cryo Cooling Collar and normothermia | 45 minutes
  Temperatures changes will be evaluated using MRI thermometry

SECONDARY OUTCOMES:
Relationship between MRI temperature of brain and externally measured temperature | 45 minutes
  Skin surface temperature probe will be used to monitor any external temperature changes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wolfson, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States